CLINICAL TRIAL: NCT05567289
Title: Precision Medicine for Stem Cell Transplantation
Acronym: PM-SCT
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mark Williams, Principal Investigator, University of Manchester
Other Study IDs: IRAS ID: 262284
Record Dates: First submitted 2022-09-28; First posted 2022-10-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-01

CONDITIONS: Haematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cryopreserved plasma and peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Blood sample collection — Enrolled patients will undergo sequential blood collection beginning prior to conditioning, then on the day of transplant (day 0), followed by days 7, 14, 21, 28, 56 (2 months) and 90 (3 months) post-transplant.
  Bone marrow aspirates taken within this period as part of routine care will also be collected, these are typically performed around day 100 and whenever there is suspicion of disease recurrence.
  The study will also collect an additional blood sample at the onset of treatment for aGvHD for those who receive systemic corticosteroids (PO or IV steroid equivalent to ≥0.5mg/kg prednisolone).
Procedure: Bone marrow aspirate — Bone marrow aspirates taken within this period as part of routine care will also be collected, these are typically performed around day 100 and whenever there is suspicion of disease recurrence.

SUMMARY:
A study of patients undergoing haematopoietic stem cell transplantation, a procedure in which patients are infused with stem cells from a donor, resulting in a new immune system that eliminates cancer or replaces diseased bone marrow. This study aims to develop new blood tests that predict the onset of acute graft-versus-host disease (aGvHD) and leukaemia relapse, two life-threatening complications that frequently limit the success of treatment. Predictive tests would allow doctors to individualise prophylaxis and intervene early to abort complications before they develop. The study will also create a large collection of clinically annotated blood samples from 300 transplant recipients to support future research and provide a resource to the transplant research community.

DETAILED DESCRIPTION:
Precision Medicine for Stem Cell Transplantation (PM-SCT) is a prospective cohort study of patients undergoing allogeneic haematopoietic stem cell transplantation (HSCT). The study aims to develop novel biomarkers that predict the onset of acute graft-versus-host disease (aGvHD) and post-transplant relapse of acute myeloid leukaemia (AML). The study will also build a collection of clinically annotated longitudinal blood samples from 300 HSCT recipients to support additional mechanistic research and provide a resource to the transplant research community.

Patients will be recruited and consented prior to admission for HSCT. Enrolled patients will undergo sequential blood collection beginning prior to conditioning, then on the day of transplant (day 0), followed by days 7, 14, 21, 28, 56 (2 months) and 90 (3 months) post-transplant. Samples will be collected, processed, and stored by the MCRC Biobank. The period of observation for each patient is 6-months. Clinical data will be collected prospectively: on admission, with each blood sample, and at 6-months post-transplant. Bone marrow aspirates taken within this period as part of routine care will also be collected, these are typically performed around day 100 and whenever there is suspicion of disease recurrence. The study aims to identify all patients who develop aGvHD, collecting an additional blood sample at the onset of treatment for those who receive systemic corticosteroids (PO or IV steroid equivalent to ≥0.5mg/kg prednisolone). Additional clinical data will be collected at treatment onset and 7, 14, 21 and 28 days after starting systemic corticosteroids. These assessments will provide the clinical data necessary to establish diagnostic confidence, severity at onset/peak, response to treatment and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Any recipient of allogeneic haematopoietic stem cell transplantation (HSCT)
* Children/infants may participate, there is no age restriction
* Patients participating in other clinical trials remain eligible

Exclusion Criteria:

* Weight <5kg
* Recipients of autologous stem cell transplants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient undergoing allogeneic haematopoietic stem cell transplantation (HSCT).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Development of biomarkers that predict the onset of acute graft-versus-host disease (aGvHD) | 5 years
  GvHD staging in this study is based on the approach of Harris et al., (2016). The weekly aGvHD assessments will provide the clinical data necessary to establish the confidence of diagnosis, severity at onset, peak severity and outcome. Four weeks of follow-up will determine whether patients achieve a complete response (CR) or very good partial response (VGPR) by day 28. In addition, the 6-month assessment will identify patients who died as a result of aGvHD and those who are alive and off immunosuppression at six months. These validated clinical endpoints will be used to identify biomarker signatures that predict aGvHD severity and response to therapy. Calendar-driven assessments will also be used to identify patients given topical steroids for grade I aGvHD as these patients may need to be excluded from use as negative controls or included as edge cases in future validation studies.

SECONDARY OUTCOMES:
Development of biomarkers that predict the relapse of acute myeloid leukaemia. | 2.5 years
  Relapse remains the leading cause of death for most transplant recipients. Approximately 40% of AML patients suffer disease recurrence, with a median time to relapse of 7 months. The 6-month follow-up assessment will therefore identify many cases of early relapse. The study will remain open for 3 years after the last assessment to allow regular updating of clinical outcome data to identify later cases of relapse. These data and the accompanying clinical samples will be used to identify cytomic and proteomic signatures of immune dysfunction and AML relapse and provide an invaluable resource for studying mechanisms of disease recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Williams, Principal Investigator — CRUK Manchester Institute
Locations (3):
- United Kingdom (3):
  - Manchester Royal Infirmary, Manchester
  - Royal Manchester Children's Hospital, Manchester
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No